CLINICAL TRIAL: NCT03605953
Title: Expansion of Invariant NKT Cells for a Cell Immunotherapeutic Approach Allowing the Control of Graft Versus Host-disease and Preserving the Graft Versus Leukemia Effect After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: ExpiNKT1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PRTK2017/ExpiNKT-RUBIO/VS
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell (HSC) Transplantation
Keywords: Cell therapy; immuno-modulation; immunotherapy; Hematology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Allogeneic hematopoietic stem cell (HSC) transplantation remains the most efficient cellular immunotherapeutic approach for the treatment of myeloid hematological malignancies. However, its use is hampered by the risk of developing acute graft-versus-host disease (aGVHD). Invariant NKT cells (iNKT) represent a good candidate of immuno-regulatory cells that could control GVHD while preserving the anti-leukemic effect (GVL) of HSCT. Our team have shown that higher numbers and expansion capacity of CD4- iNKT cells contained in the HSC graft were associated with reduced risk of aGVHD but preserved GVL effect and that some healthy donors have low numbers and expansion capacity CD4- iNKT cells 1.

The objective of this project is to develop a strategy allowing to expand human CD4- iNKT cells from healthy donors of HSC grafts that would be transposable to GMP-validated cell production. Our team proposes to first determine the best strategy to expand the CD4- iNKT cell subset from G-SCF mobilized peripheral blood stem cells (PBSC) obtained from healthy donors, at little scale using cultures GMP validated conditions, by comparing the convention expansion protocol using IL-2 alone to IL-7, IL-15, IL-4 or combination of those cytokines involved in the expansion of T cells and by culturing the cells in a bioreactor. Our team will then explore the characteristics of cells after expansion in terms of phenotype, transcription signature and functions in vitro (in mixed lymphocyte reaction) and in vivo in a well-established xenogeneic model of GVHD.

ELIGIBILITY:
Inclusion Criteria:

Hematopoietic stem cells :

* from major donors after mobilization by G-CSF, informed of the research and not having opposed it
* Collected after verification by the cell therapy centre of the presence of a sufficient quantity of CSH for transplantation

Exclusion Criteria:

Hematopoietic stem cells (HSCs) from donors seropositive for HIV, HCV, HTLV1 and HBV (except post-vaccination profile)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: healthy donors of HSCT
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Kinetic of iNKT cells (flask culture) | from day 0 to day 14
time of culture to reach the maximal expansion factor | day 14
Percentage of cells alive | day 14
Percentages of CD4- iNKT cells capable of producing IFN-γ after expansion | day 14

SECONDARY OUTCOMES:
Kinetic of iNKT cells(culture in bioreactor system) | From day 0 to day 14
Expression of cytokine receptors CD4- iNKT data | day 14
Expression of cytokine receptors CD4+ iNKT data | day 14
transcriptional pattern CD4- iNKT data | day 14
Transcriptional pattern CD4+ iNKT | day 14
Percentage of recovery of CD4- iNKT cells after immunomagnetic selection | day 14
Proportion of Th1 producing T cells stimulated by allogeneic dendritic cells | day 6 in a mixed lymphocyte reaction
Proportion of Th17 producing T cells stimulated by allogeneic dendritic cells | day 6 in a mixed lymphocyte reaction
Proportion of mice protected from GVHD mortality in a xeno-GVHD mouse model | survival proportions between day 28 and day 60 post-transplantation
Ratio of iNKT/T cells to control xeno-GVHD mortality | survival proportions between day 28 and day 60 post-transplantation
Proportion of mice protected from leukemia development | survival proportions between day 28 and day 60 post-transplantation